CLINICAL TRIAL: NCT04692467
Title: Treatment of Early Hypertension Among Persons Living With HIV in Haiti
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-03021735; R21TW011693 (NIH)
Record Dates: First submitted 2020-12-15; First posted 2020-12-31 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: HIV/AIDS; Pre Hypertension
Keywords: hypertension; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Prehypertension; Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Early hypertension) (Experimental): Participants randomized to the early HTN treatment arm will initiate 5mg daily of amlodipine immediately, increasing to 10 mg if SBP >130 mmHg after 1 month.
  Interventions: Drug: Amlodipine 5mg
- Standard of Care (No Intervention): Participants randomized to the SOC arm will not be initiated on any medications initially. They may be initiated on amlodipine only if they develop HTN (SBP ≥140 or DBP ≥90 mm Hg).

INTERVENTIONS:
Drug: Amlodipine 5mg — Amlodipine, Haiti's first-line antihypertensive medication, will be administered to the intervention group.
  Other Names: Norvasc
  Arms: Intervention (Early hypertension)

SUMMARY:
The investigators are conducting an unblinded pilot randomized control trial of 250 persons living with HIV (PLWH), aged 18-65 years, who receive antiretroviral therapy care at Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic Infections (GHESKIO), are virally suppressed, and have pre-hypertension (systolic blood pressure (SBP) 120-139 or diastolic blood pressure (DBP) 80-89 mmHg) to be randomized to early hypertension (HTN) treatment versus standard of care (SOC). Participants will be recruited from GHESKIO's HIV clinic. Eligible individuals will complete informed consent and be randomized to early HTN treatment vs. SOC. Participants in early HTN treatment will initiate amlodipine immediately versus those in SOC will initiate amlodipine only if they meet the HTN threshold (SBP ≥140 or DBP ≥90 mmHg) during the study period. All participants will be followed for 12 months.

DETAILED DESCRIPTION:
The investigators propose a pilot randomized controlled trial to evaluate antihypertensive treatment among people living with HIV (PLWH) with pre-hypertension (pre-HTN) at GHESKIO. This study will provide critical data on the feasibility, benefits and risks of antihypertensive treatment for cardiovascular disease (CVD) prevention among PLWH with pre-HTN that will inform a future definitive trial powered for incident CVD events.

For the pilot study, the investigators will enroll 250 PLWH (18-65 years of age) who have been on antiretroviral therapy (ART) for ≥ 1 years with viral suppression within past 12 months and SBP 120-139 or DBP 80-89 mm Hg and no current antihypertensive treatment; randomize them to "early HTN treatment" or the current standard of care (SOC); and follow them for 12 months. Amlodipine is the recommended first-line anti-hypertensive medication according to Haiti's new primary care HTN guidelines. Participants in the early HTN treatment arm will initiate amlodipine 5 mg immediately, increasing to 10 mg if SBP >130 mm Hg after 1 month. Participants in the SOC arm will initiate amlodipine only if they develop HTN (SBP ≥140 or DBP ≥90 mm Hg).

Participants that meet study eligibility criteria will proceed to study enrollment visit (~90 min). Participants will be randomized to early HTN treatment vs. SOC in a 1:1 ratio using a computer-generated random assignment. The research nurse will collect demographic and clinical data, administer a baseline questionnaire, measure unobserved BP, and perform an ECG. The questionnaire includes a CVD medical history, family history, medications, CVD health behaviors (smoking, alcohol, physical activity, and diet) using validated questions that have been used at GHESKIO and are comparable to those used in US cohorts. Enrollment labs (~15ml of venous blood) including HgbA1c, total cholesterol, high density cholesterol, CD4 (cluster of differentiation 4) cell count, and HIV viral load (unless available from electronic medical record in the past 6 months) will be collected. Samples of serum and plasma will be stored for future studies, with documented consent from participants. The study physician will interpret the ECG and perform an echocardiogram and vascular ultrasound.

Study drug will be dispensed to participants randomized to the early treatment arm with appropriate education and counseling on adherence and potential side effects. Amlodipine will be started at 5mg at enrollment and increased to 10mg if SBP >130 mm Hg after 1 month for participants in the early treatment arm. Locator and contact information will be verified and follow up appointment given.

After enrollment and randomization assignment (including amlodipine initiation), participants will have follow-up visits either at GHESKIO (months 0.5-1, 3, 6, 9, 12) or in the community / home with community health workers (months 2, 5, 8). All visits will include BP measurement, lifestyle counseling, adherence encouragement, and assessment of adverse events. The GHESKIO visits will also include a physical exam. Participants in the early intervention arm will receive monthly amlodipine refills. Participants in the SOC arm will initiate amlodipine only if they develop hypertension (SBP >140 or DBP >90 mm Hg).

At the 12-month study visit, participants will also complete a brief questionnaire about changes in health behaviors and have viral load measured. Participants may return to the HIV clinic at any time for symptoms, questions, or other concerns, and a BP measurement will be taken at each of these encounters. Adverse events will be assessed at each visit. Medical record abstraction will be done by research staff for any hospitalization or death among a participant.

ELIGIBILITY:
Inclusion Criteria:

* PLWH 18-65 years of age
* ART duration ≥ 1 year, stable regimen ≥ 6 months
* HIV 1-RNA < 1,000 copies/mL within past 12 months
* Pre-HTN (SBP 120-139 or DBP 80-89 mm Hg)
* No current antihypertensive treatment
* Receives HIV care at GHESKIO
* Willing to provide consent

Exclusion Criteria:

* Pregnancy
* Kidney disease or diabetes
* On protease inhibitor/ritonavir
* Advanced illness with limited life expectancy
* Plans to move out of the area within the next year
* Clinician determination that patient is unstable on ART

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNairy, MD, Principal Investigator — Weill Medical College of Cornell University; Jean Pape, Principal Investigator — Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic
Locations (1):
- GHESKIO, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data collected during the trial, after deidentification will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and statistical analysis plan available after publication and ending 3 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal may have access. Proposals should be directed to the PI at mam9365@med.cornell.edu. To gain access, data requestors will need to sign a data access agreement. Data are available following publications through 3 years after publication and will be provided directly from the PI.

REFERENCES:
- [Derived] Yan LD, Rouzier V, Sufra R, Sauveur RS, Guiteau C, Lee MH, Ogyu A, Mourra N, Oparil S, Theard M, Brisma JP, Alfred JP, Deschamps MD, Pape JW, McNairy ML. Treatment of prehypertension among adults with HIV. AIDS. 2025 Mar 1;39(3):261-269. doi: 10.1097/QAD.0000000000004065. Epub 2024 Nov 13. PMID 39761592
- [Derived] Yan LD, Rouzier V, Dade E, Guiteau C, Pierre JL, St-Preux S, Metz M, Oparil S, Pape JW, McNairy M. Treatment of early hypertension among persons living with HIV in Haiti: Protocol for a randomized controlled trial. PLoS One. 2021 Aug 5;16(8):e0254740. doi: 10.1371/journal.pone.0254740. eCollection 2021. PMID 34351939

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Started | 124 | 126
Completed | 124 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: In intention-to-treat analysis, the analysis population is the same as the assignment under randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (Early Hypertension) | Standard of Care | Total
Number analyzed (Participants) | 124 | 126 | 250
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.0 [48.3 to 55.3] | 47.5 [41.3 to 55.0] | 49.0 [42.0 to 55.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 54 | 102
  Male | 76 | 72 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 124 | 126 | 250
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 124 | 126 | 250
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Haiti | 124 | 126 | 250
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 129 [126 to 132] | 128 [126 to 133] | 129 [126 to 132]

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Systolic Blood Pressure (SBP)
Time Frame: Baseline, 12 months
Population: For participants receiving Standard of Care, 120 of the 126 (95.2%) had a 12-month visit. For the participants receiving the intervention, 122 of the 124 (98.4%) had a 12-month visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
mmHg | -10.58 (11.01) | -4.65 (11.41)
Statistical Analysis 1: Comparison: Intervention (Early Hypertension) vs Standard of Care; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -5.88, 95% CI 2-sided [-8.77 to -3.01] — The mean difference reflects the difference in mean change (i.e., mean change = 12 months minus baseline for each arm) between the intervention arm and SOC arm (direction = intervention arm minus SOC arm)

2. Secondary Outcome: Change in Number of Participants With HIV Viral Suppression as Measured by HIV-1 RNA Viral Loads < 1,000 Copies/mL
Time Frame: Baseline, 12 months
Population: At the 12-month visit, 8 participants in the Standard of Care arm and 5 participants in the intervention arm were missing viral load data.
Measure: Number; unit: participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
participants
  Baseline | 124 | 126
  12 months | 115 | 114

3. Secondary Outcome: Change in HIV Medication Adherence as Measured by Number of Participants With > 90% Adherence Using 4-day Pill Recalls
Time Frame: Baseline, 6 months and 12 months
Measure: Number; unit: participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
participants
  Baseline | 107 | 114
  6 months | 98 | 91
  12 months | 111 | 99

4. Secondary Outcome: Number of Subjects Who Have Adverse Events Related to Amlodipine, Including Dizziness, Fainting, Lower Extremity Edema, and Any Other Symptoms Which May be Related.
Description: Symptoms will be categorized according to the Division of AIDS (DAIDS) severity score, with Grade III-IV considered adverse events.
Time Frame: Followup month 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
Participants | 10 | 0

5. Secondary Outcome: Number of Subjects Who Have Adverse Events Related to Amlodipine, Including Dizziness, Fainting, Lower Extremity Edema, and Any Other Symptoms Which May be Related.
Description: as for outcome 4
Time Frame: Followup month 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
Participants | 8 | 0

6. Secondary Outcome: Number of Subjects Who Have Adverse Events Related to Amlodipine, Including Dizziness, Fainting, Lower Extremity Edema, and Any Other Symptoms Which May be Related.
Description: as for outcome 4
Time Frame: Followup month 3
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
Participants | 0 | 0

7. Secondary Outcome: Adverse Events
Description: Number of subjects who have adverse events related to amlodipine, including dizziness, fainting, lower extremity edema, and any other symptoms which may be related. Symptoms will be categorized according to the Division of AIDS (DAIDS) severity score, with Grade III-IV considered adverse events.
Time Frame: Followup month 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
Participants | 3 | 0

8. Secondary Outcome: Number of Subjects Who Have Adverse Events Related to Amlodipine, Including Dizziness, Fainting, Lower Extremity Edema, and Any Other Symptoms Which May be Related.
Description: as for outcome 4
Time Frame: Followup month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
Participants | 2 | 0

9. Secondary Outcome: Number of Subjects Who Have Adverse Events Related to Amlodipine, Including Dizziness, Fainting, Lower Extremity Edema, and Any Other Symptoms Which May be Related.
Description: as for outcome 4
Time Frame: Followup month 8
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 126
Participants | 1 | 0

10. Secondary Outcome: Number of Subjects Who Have Adverse Events Related to Amlodipine, Including Dizziness, Fainting, Lower Extremity Edema, and Any Other Symptoms Which May be Related.
Description: as for outcome 4
Time Frame: Followup month 9
Population: 1 participant in the standard of care arm was excluded from analysis because the participant died of causes unrelated to the research prior to follow-up month 9.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 125
Participants | 0 | 0

11. Secondary Outcome: Number of Subjects Who Have Adverse Events Related to Amlodipine, Including Dizziness, Fainting, Lower Extremity Edema, and Any Other Symptoms Which May be Related.
Description: as for outcome 4
Time Frame: Followup month 12
Population: 2 participants in the standard of care arm were excluded from analysis because these participants died of causes unrelated to the research prior to follow-up month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 124
Participants | 0 | 0

12. Secondary Outcome: Number of Participants Who Are Enrolled at Baseline and Remain in the Study by 12 Months
Description: All participants were included in enrolment. Remaining in the study was defined as having a clinic visit at month 12 (final study visit).
Time Frame: Baseline, 12 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Early Hypertension) | Standard of Care
Number analyzed (Participants) | 124 | 124
Participants | 122 | 120

13. Secondary Outcome: Acceptability of Study Intervention Assessed by Qualitative Interviews Among Participants and Providers
Description: Using semi-structured interview guides exploring topics including acceptability, side effects, perceived benefit, and perceived cost, in depth interviews will be conducted with 15-20 study participants in the intervention arm, and all healthcare providers involved in the study (nurses, doctors, social workers).
Time Frame: 12 months
Population: Focus-group discussions were conducted with participants who received the intervention. A subset of 16 participants were randomly selected and called to conduct FGD. Individual interviews were conducted with providers. All physicians (two) who were involved in the study were interviewed. One nurse was excluded as they could not be contacted as they had left the clinic.
Measure: Number; unit: participants
Groups:
- Intervention (Early Hypertension): Patients who participated in the study who were given the intervention were invited to a focus-group discussion. In each session there were 6-8 participants.
- Providers: Providers who were part of the study and also consented to being interviewed
Arm/Group | Intervention (Early Hypertension) | Providers
Number analyzed (Participants) | 16 | 2
participants
  Satisfaction | 8 | 2
  Positive Effects | 12 | 2
  Negative Effects | 10 | 2
  Intent to continue | 11 | 0
  Amlodipine Initiation | 3 | 2
  CVD Risk | 10 | 2
  Unintended consequences | 0 | 2
  Implementation Challenges | 6 | 2

ADVERSE EVENTS:
Time Frame: All participants were asked at each community and clinic visit whether they had adverse events. Clinic visits occurred at 1, 3, 6, 9, and 12 months after enrolment. Community visits occurred at 2, 5, and 8 months after enrolment. Participants were followed up for up to 12 months after enrollment.
Description: Signs and symptoms of hypotension and peripheral edema, or any other reported side effects were graded using the existing Division of AIDS (DAIDS) criteria.
Arm/Group | Intervention (Early Hypertension) | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/124 | 2/126
Serious Adverse Events (participants affected / at risk) | 1/124 | 0/126
Other Adverse Events (participants affected / at risk) | 22/124 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (Early Hypertension) (N=124) | Standard of Care (N=126)
Marked weakness (General disorders) | 1 (1) | 0 (0) — Grade 3: severe
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (Early Hypertension) (N=124) | Standard of Care (N=126)
Edema (Cardiac disorders) | 4 (4) | 0 (0) — Grade 1: mild
Edema (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2: moderate
Fatigue (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2: moderate
Headache (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2: moderate
Dizziness (Cardiac disorders) | 12 (12) | 0 (0) — Grade 1: mild
Dizziness (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2: moderate
Urine Flow Increase (Renal and urinary disorders) | 2 (2) | 0 (0) — Grade 1: mild
Neck Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 2: moderate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04692467/Prot_SAP_001.pdf